CLINICAL TRIAL: NCT01233115
Title: LOC387715/HTRA1 Variants and the Response to Combined Photodynamic Therapy With Intravitreal Bevacizumab in Polypoidal Choroidal Vasculopathy
Brief Title: LOC387715/HTRA1 and the Combined Photodynamic Therapy With Intravitreal Bevacizumab in Polypoidal Choroidal Vasculopathy
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, clinical professor, Kyungpook National University Hospital
Other Study IDs: LOC387715/HTRA1 & combined PDT
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Genomic DNA was extracted from peripheral blood. The two SNPs (rs10490924 in the LOC387715 locus and rs11200638 in HTRA1 gene) were analyzed by LC480 Real time PCR (Roche, Basel, Switzerland) at D&P Biotech (Daegu, Korea).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- polypoidal choroidal vasculopathy: patients who were treated for polypoidal choroidal vasculopathy with combined photodynamic therapy and intravitreal bevacizumab injections

SUMMARY:
This study is to investigate whether there is an association of the LOC387715/HTRA1 variants with response to treatment with combined photodynamic therapy and intravitreal bevacizumab for patients with polypoidal choroidal vasculopathy.

DETAILED DESCRIPTION:
This is a retrospective cohort study comprised of 70 eyes being treated for polypoidal choroidal vasculopathy with combined photodynamic therapy and intravitreal bevacizumab injections. Patients were genotyped for the LOC387715 (rs10490924) and the HTRA1 gene polymorphism (rs11200638).

ELIGIBILITY:
Inclusion Criteria:

* patients older than 60 years of age at onset
* polyp-like terminal aneurysmal dilations with or without branching vascular networks in indocyanine green angiography (ICGA) and subretinal reddish-orange protrusions corresponding to polyp-like lesions
* patients who had combined photodynamic therapy and intravitreal bevacizumab injections, and followed up for more than 12 months after the first treatment

Exclusion Criteria:

* patients with retinal or choroidal diseases including pathologic myopia, angioid streaks, idiopathic choroidal neovascularization (CNV), presumed ocular histoplasmosis, and other secondary CNV
* patients who refused genotypic analyses

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The authors did a retrospective chart review of 70 patients with PCV who were treated at the Department of Ophthalmology, Kyungpook National University Hospital in Daegu, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | up to 12 months
  Best-corrected visual acuity (BCVA) using the Snellen chart was evaluated including BCVA up to 12 months

SECONDARY OUTCOMES:
Angiographic characteristics | up to 12 months
  Fluorescein angiography (FA) and ICGA (HRA; Heidelberg Engineering, Dossenheim, Germany) was evaluated. Greatest linear dimension (GLD) was determined based on both FA and ICGA.

CONTACTS AND LOCATIONS:
Overall Officials: In Taek Kim, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- In Taek Kim, Daegu, Kyungsangpookdo, South Korea

REFERENCES:
- [Result] Sakurada Y, Kubota T, Imasawa M, Mabuchi F, Tanabe N, Iijima H. Association of LOC387715 A69S genotype with visual prognosis after photodynamic therapy for polypoidal choroidal vasculopathy. Retina. 2010 Nov-Dec;30(10):1616-21. doi: 10.1097/IAE.0b013e3181e587e3. PMID 20671585
- See also: genetics home reference — http://ghr.nlm.nih.gov/